CLINICAL TRIAL: NCT00992030
Title: Phase III Study Comparing Rituximab-supplemented ABVD (R-ABVD) With ABVD Followed by Involved-field Radiotherapy (ABVD-RT) in Limited Stage (Stage I-IIA With no Areas of Bulk) Hodgkin's Lymphoma
Brief Title: R-ABVD vs ABVD-RT in Early Stage Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment and difficulty in having study data
Sponsor: Fondazione Michelangelo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-HD09-01; 2009-009431-30 (EudraCT Number)
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2019-07

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Rituximab; ABVD protocol; Bleomycin; Vinblastine; Dacarbazine; Doxorubicin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Experimental): Rituximab plus ABVD (doxorubicin, bleomycin, vinblastine, dacarbazine) for 4 cycles
  Interventions: Drug: Rituximab
- ARM B (Active Comparator): ABVD (doxorubicin, bleomycin, vinblastine, dacarbazine) for 4 cycles followed by involved field irradiation
  Interventions: Radiation: Involved field irradiation

INTERVENTIONS:
Drug: Rituximab — I.V. infusion weekly x 6 weeks at a dose of 375 mg/m2
  Other Names: Drug: rituximab; Drug: ABVD regimen; Drug: doxorubicin hydrocloride; Drug: bleomycin; Drug: vinblastine; Drug: dacarbazine
  Arms: ARM A
Radiation: Involved field irradiation — Radiation therapy, limited to initially involved nodal sites, will start within four weeks from the last cycle of ABVD chemotherapy and after complete restaging with TAC total-body and PET total-body. The planned total dose is 30,6 Gy.
  Other Names: Drug: ABVD regimen; Drug: doxorubicin hydrochloride; Drug: bleomycin; Drug: vinblastine; Drug: dacarbazine; Radiation: radiation therapy
  Arms: ARM B

SUMMARY:
Combined modality therapy has then emerged as the standard of care for limited-stage Hodgkin's lymphoma and doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) chemotherapy that is devoid of alkylating agents and associated with a low potential for gonadal toxicity and leukemogenesis, is currently considered a gold standard. Nevertheless, the disadvantage to combine radiotherapy to ABVD is represented by late cardiovascular events (myocardial dysfunction and coronary or valvular disease), especially when the heart is within the radiation field; bleomycin pulmonary toxicity also is increased in conjunction with RT and secondary tumors, in particular in the RT fields. This study aims at treating patients with limited disease with multiagent chemotherapy alone, without irradiation, and using radiotherapy only for relapses.

DETAILED DESCRIPTION:
Limited-stage Hodgkin lymphoma is a highly curable disease, with expected long-term disease-free and overall survival rates close to 90% and 95%, respectively. This success has come at a cost of long-term treatment-related toxicity, such that the patients who live beyond 10 to 15 years are more likely to die from late complications of treatment than from the disease itself. In the last decades efforts to improve long-term results have been made by developing curative strategies aimed to reduce toxicity while maintaining high cure rates. Based on the observation that systemic chemotherapy can control occult sites of the disease, thereby eliminating the requirement for staging laparotomy, in the last years the use of combined modalities that allowed a reduction of number of cycles of chemotherapy and of radiation field size and doses, thus reducing late toxicity was investigated in various clinical trials. Combined modality therapy has then emerged as the standard of care for limited-stage Hodgkin's lymphoma and doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) chemotherapy that is devoid of alkylating agents and associated with a low potential for gonadal toxicity and leukemogenesis, is currently considered the gold standard. Nevertheless, optimal treatment is still a question of debate and current investigations are now taking into consideration to further reduce long-term toxicity. Actually two main options are available. The first option combines radiotherapy to ABVD chemotherapy, with the aim to maximize disease control. Using 4 cycles of ABVD followed by involved field radiotherapy at 36 Gy, Bonadonna and coworkers first documented a 94% freedom-from-progression and a 94% overall survival rate, respectively. The disadvantage with this approach is represented by late cardiovascular events (myocardial dysfunction and coronary or valvular disease), especially when the heart is within the radiation field; bleomycin pulmonary toxicity also is increased in conjunction with RT and secondary tumors, in particular in the RT fields. Whether these risks will be lower with fewer chemotherapy cycles, lower RT doses, or both has been studied in many clinical trials that have demonstrated that smaller radiation fields and lower doses are important, but a key unanswered question is whether RT can be eliminated completely in limited-stage patients. The second option therefore consists of chemotherapy with ABVD alone, with the aim to eliminate the late effects of radiotherapy. This approach have resulted in an absolute increase of the failure rate in the order of 8% (from approximately 4% up to 12%). However, the majority of relapsing patients achieves a durable disease control with a second-line radiation-containing combined approach, and shows an overall survival rate superimposable to that of patients receiving upfront combined strategy with chemo-radiotherapy. We thus designed a study aimed at treating patients with limited disease with multiagent chemotherapy alone, without irradiation, and using radiotherapy only for relapses. In fact, it has recently been reported that the addition of Rituximab (a monoclonal antibody directed against the CD20 B-cell antigens) to ABVD significantly increases the antilymphoma activity of ABVD alone in advanced-stage Hodgkin's lymphoma and in absence of added toxicity. In conclusion, rituximab-supplemented ABVD (R-ABVD) given to early-stage Hodgkin's lymphoma might represent a radiation-free regimen capable of increasing long-term disease control of ABVD alone, while avoiding the late effects of radiotherapy.

The primary objective of this study is to evaluate whether the R-ABVD therapy (ARM A) is not worse than the standard therapy of ABVD-RT (ARM B) in patients with limited Hodgkin's lymphoma. In this trial a maximum inferiority of 8% of the 3-year Failure Free Survival rate (FFS) in ARM A with respect to ARM B is considered acceptable to assess that ARM A is not worse than ARM B.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed classical Hodgkin lymphoma (cHL)
* Limited-stage disease defined as stage I or IIA with no areas of bulky disease
* Measurable disease according to the Cheson criteria
* Age >=18 years
* Adequate bone marrow reserve (ANC >= 1,500/uL, Platelet > 100,000/uL)
* LVEF >= 50% by MUGA scan or echocardiogram
* Serum creatinine < 2 mg/dl, serum bilirubin < 2 mg/dl, AST or ALT <2x ULN
* Bi-dimensionally measurable disease
* Use of effective means of contraception
* Signed informed consent form

Exclusion Criteria:

* Lymphocyte predominant HL
* Prior chemotherapy or radiation therapy
* Severe pulmonary disease as judged by the PI including COPD and asthma
* Presence of CNS lymphoma
* Concomitant malignancies or previous malignancies (exception made for adequately treated basal or squamous cell carcinoma of the skin)
* Active infection requiring treatment with intravenous therapy
* Known HIV infection
* Active hepatitis B or C
* Pregnancy or lactation and women of child bearing age who are not practicing adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-09; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
3-year failure free survival. Failure is defined as disease progression during treatment, achievement of less than complete remission (CR) after the total planned therapy, relapse during follow-up or death from any cause. | Three-year failure free survival from randomization

SECONDARY OUTCOMES:
Event-free survival including, besides failures, late serious treatment-related events | 7 years from randomization
Overall survival, all causes included | 7 year from randomozation

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro M Gianni, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (11):
- UT MD Anderson Cancer Center, Houston, Texas, United States
- Italy (10):
  - Ospedali Riuniti Umberto I, Ancona
  - Ospedali Riuniti, Bergamo
  - Policlinico S. Orsola Malpighi, Bologna
  - Ospedale Roberto Binaghi, Cagliari
  - Azienda Ospedaliera Vittorio Emanuele Ferrarotto, Catania
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Azienda Ospedaliero Universitaria S. Luigi Gonzaga, Orbassano
  - Gianpietro Semenzato, Padua
  - Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Ospedale San Carlo, Potenza